CLINICAL TRIAL: NCT05344157
Title: A First-in-Human Open-Label Phase 1/2a Study to Evaluate Safety, Tolerability and Efficacy of a Single Intra-Articular Injection of Allogeneic Mesenchymal Stem Cells Selected for Integrin α10β1 (XSTEM-OA) in Adult Patients With Symptomatic Knee Osteoarthritis
Brief Title: A First-in-Human Study of XSTEM-OA in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xindu Pty Ltd (Industry)
Collaborators: Xintela AB (Industry)
Responsible Party: Sponsor
Organization: Xintela AB (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XIN-XSTEM-101
Record Dates: First submitted 2022-04-04; First posted 2022-04-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XSTEM-OA (Experimental): Single intra-articular injection of XSTEM-OA
  Interventions: Biological: XSTEM-OA

INTERVENTIONS:
Biological: XSTEM-OA — XSTEM-OA is an allogeneic, adipose tissue-derived, integrin alpha10beta1-selected and expanded mesenchymal stem cell (MSC) product for the treatment of osteoarthritis.

SUMMARY:
The aim of the study is to assess safety, tolerability and preliminary efficacy of XSTEM-OA when administered as a single intra-articular injection to patients with symptomatic knee osteoarthritis. The study is divided into two parts; a dose escalation (Part A) and an optional dose expansion part (Part: B). Three dose levels are planned to be evaluated in Part A and selected dose level(s) may be further expanded in Part B.

ELIGIBILITY:
Major inclusion criteria:

* Aged ≥40 and ≤75 years at Screening
* Radiological evidence of predominantly medial osteoarthritis in the knee, uni- or bilateral, of KL grade II to III
* Moderate to severe pain associated with osteoarthritis in the knee as measured by a VAS pain score of ≥35 and ≤90 mm

Major exclusion criteria:

* Body mass index (BMI) of ≥35 at Screening
* Ongoing signs or symptoms of systemic or local infection
* Known knee infection in the study knee within 6 months of Screening
* History of clinically relevant concomitant joint disease, clinically-relevant knee deformities, or any clinically significant medical history of the ligament, or realignment surgery or joint replacement surgery
* Medical history of any autoimmune disease
* History of surgery in the study knee that occured within 6 months of Screening
* Treatment with immunosuppressive therapy (systemic or local) or any medication affecting the bone or cartilage metabolism within 6 months of Screening
* Patients who are immunocompromised as caused by a disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AEs) | From start of study until 24 months after injection
  Incidence, nature and severity of treatment-related AEs assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Safety and tolerability: 12-lead electrocardiogram (ECG) | From start of study until 18 months after injection
  Change in 12-lead electrocardiograms (ECGs) compared to baseline.
Safety and tolerability: Laboratory examinations | From start of study until 18 months after injection
  Changes in laboratory tests compared to baseline. The clinical laboratory tests include haematology, chemistry, coagulation and urinalysis.
Safety and tolerability: Physical examinations | From start of study until 18 months after injection
  Changes in physical examination compared to baseline.
Safety and tolerability: Vital signs | From start of study until 18 months after injection
  Changes in vital signs compared to baseline. Vital signs include blood pressure, pulse rate, respiratory rate and oral body temperature.

SECONDARY OUTCOMES:
Preliminary efficacy: Changes in Visual Analogue Scale (VAS) for pain compared to baseline | From start of study until 18 months after injection
Preliminary efficacy: Changes in Knee injury and Osteoarthritis Outcome Score (KOOS) compared to baseline | From start of study until 18 months after injection
Preliminary efficacy: Change in EuroQoL 5 Dimension 5 Level test (EQ-5D-5L) compared to baseline | From start of study until 18 months after injection
Preliminary efficacy: Change in 40 m fast paced walk test compared to baseline | From start of study until 18 months after injection
Preliminary efficacy: Change in cartilage structure and morphology compared to baseline, based on MRI assessment of cartilage volume and composition | From start of study until 18 months after injection
Preliminary efficacy: Change in whole knee health compared to baseline, based on MRI assessment by the MRI Osteoarthritis Knee Score (MOAKS) | From start of study until 18 months after injection
Preliminary efficacy: Change in inflammatory activity compared to baseline, based on MRI assessment of synovitis | From start of study until 18 months after injection
Preliminary efficacy: Changes in joint space narrowing based on x-ray compared to baseline | From start of study until 18 months after injection

OTHER OUTCOMES:
Exploratory outcome: Change in Visual Analogue Scale (VAS) for pain compared to baseline | 24 months after injection
Exploratory outcome: Change in KOOS compared to baseline | 24 months after injection
Exploratory outcome: Change in EQ-5D-5L compared to baseline | 24 months after injection
Exploratory outcome: Change in 40 m fast paced walk test compared to baseline | 24 months after injection
Exploratory outcome: Change in cartilage structure and morphology compared to baseline, based on MRI assessment of cartilage volume and composition | 24 months after injection
Exploratory outcome: Change in whole knee health compared to baseline, based on MRI | 24 months after injection
Exploratory outcome: Change in inflammatory activity compared to baseline, based on MRI assessment of synovitis | 24 months after injection
Exploratory outcome: Change in joint space narrowing based on x-ray compared to baseline | 24 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Per Norlén, MD, PhD, Study Director — Xintela AB; Stephen Hall, Dr, Principal Investigator — Emeritus Research
Locations (2):
- Australia (2):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Emeritus Research, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No